CLINICAL TRIAL: NCT01920529
Title: Effectiveness of a Physical Training Program on Inflammatory Response, Functional Capacity and Quality Life in Children With Moderate and Severe Asthma.
Brief Title: Aerobic Exercise in Children With Moderate and Severe Asthma
Acronym: AECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Livia Barboza de Andrade, PhD Student, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: livia1971; EASMADOC2013 (Other: University Hospital)
Record Dates: First submitted 2013-05-13; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: asthma, aerobic exercise, child, cytokines
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic exercise (Experimental): The study will consist of two groups: Group Comparison (GC) will be submitted to two evaluations at the beginning of a week and end of 6 weeks, without receiving any kind of physical training intervention. Group Training (GT) will undergo two assessments at the beginning of the end of the 1st and 6th week, however will be submitted to aerobic training for six weeks. Supervised aerobic training will be held three times a week for six weeks,treadmill in four consecutive steps each (05 minutes stretching, 05 minutes heating, 20 training minutes (1 st and 2 nd week) and 30 minutes (3 rd to 6 weeks) and cool down 05 minutes). The exercise intensity will be maintained through a desired percentage of heart rate for training (x%) from 70% to 80%, obtaining then the optimal heart rate training.
  Interventions: Other: aerobic exercise
- control (Placebo Comparator): Investigators evaluated the distance walked during the 6-minute walk test and recorded variables such as heart rate, respiratory frequency, pulse oxygen saturation and a scale of perceived exertion (Borg) in the moments before and after the test. There was only evaluation without intervention.
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — Performed aerobic exercise on a treadmill with cardiac predetermined frequency within 6 weeks and frequency of three times per week. All patients were monitored during training.
  Other Names: physical exercise, physical training

SUMMARY:
Regular aerobic physical activity in short-term moderate asthma and severe:

* Reduce the levels of inflammatory mediators
* Improves functional capacity
* Improves Quality of Life
* Improved lung function
* Reduces the sensation of dyspnea
* Improves symptoms scores and medication use

DETAILED DESCRIPTION:
Methods: Is designed a randomized clinical trial, efficacy, outpatient physical therapy developed in the Institute of Integrative Medicine Teacher Fernando Figueira (IMIP). A pilot study with 20 participants will be made initially to obtain a sample calculation. Subjectively estimated it will take about 50 participants, with possible losses. Will include children older than eight years, diagnosis of moderate and severe persistent asthma according to criteria of Global Initiative National Asthma (GINA) and forced expiratory volume in one minute (FEV1) below 80% predicted. Will be excluded from the study associated with disease that limits physical activity, such as neuromuscular diseases, congenital or acquired heart disease, chronic lung disease associated exacerbation of the crisis and significant cognitive deficit, which makes the participant to respond adequately to the questionnaire and / or inability to meet the commands. Eligible patients will be randomized into two groups: control group, which is not subjected to any kind of exercise and the intervention group, which will be submitted to aerobic exercise for 30 minutes three times a week for six weeks. The two groups will be evaluated before and at the end of six weeks by testing for 6-minute walk, analysis of dyspnea, questionnaire of quality of life, pulmonary function test (FEV1, FVC), inflammatory markers (cytokine ).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than eight and less than nineteen years
* Diagnosis of moderate to severe persistent asthma according to criteria of GINA
* forced expiratory volume in one minute (FEV1) below 80% of predicts
* Initiation of treatment with inhaled corticosteroids for at least eight weeks before the start of collection.

Exclusion Criteria:

* associated disease that limits physical activity, such as neuromuscular disease, congenital or acquired, severe cor pulmonate, severe congenital malformation
* associated with chronic lung disease (cystic fibrosis, bronchiectasis, bronchopulmonary dysplasia, interstitial lung diseases
* significant cognitive deficit, which makes the participant to respond adequately to the questionnaire and / or failure to meet the commands
* exacerbation of crisis (This will be a temporary exclusion criterion, as having taken action as directed by medical routine, the participant can return to training)
* mental deficit.

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory mediators by analyzing cytokines by flow cytometry | six weeks
  Was carried collection of peripheral blood cells separated and analyzed for cytokine flow cytometry method. We evaluated Th1 and Th2 cytokines.

SECONDARY OUTCOMES:
Distance walked during the 6-minute walk | 6 weeks
  Before and after 6 weeks of intervention
Changes in lung function | Before and after 6 weeks of intervention
  Assessed by spirometry (forced expiratory volume in one second, forced vital capacity and the relationship of these. Besides, peak expiratory flow.
Days free of asthma | After six weeks
  Measured through a journal that will be recorded days without asthma symptoms such as cough, dyspnea, chest tightness, and use of extra medication.
Respiratory pressures maxima | Before and after 6 weeks
  Through the evaluation of the maximum inspiratory and expiratory pressure by manuvacuometro
Analysis of cytokines | Before and after 6 weeks
  Measured in blood plasma samples and analyzed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Livia B Andrade, PhD student, Principal Investigator — Professor of Pediatric Physical Therapy Specialization of integral medicine institute Prof. Fernando Figueira
Locations (1):
- Integral Medicine Institute Professor. Fernando Figueira-IMIP, Recife, Pernambuco, Brazil